CLINICAL TRIAL: NCT06561191
Title: Effects of Dialyzer Characteristics and Dialysis Mode on Functional Properties of Albumin in Patients With Chronic Hemodialysis Treatment
Brief Title: Functionality of Albumin in the Context of Hemodialysis
Acronym: FACED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Kristina Boss, PD Dr. med. Kristina Boss, Universität Duisburg-Essen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024_EKEA.29
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Albumin; Dialysis; Redox State; Uremic; Toxemia
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): All patients recieve three month of treatment with hemodialysis, hemodiafiltraten, treatment with high flux dialyzer and treatment with low flux dialyzer
  Interventions: Other: Hemodialysis mode, dialyzer type

INTERVENTIONS:
Other: Hemodialysis mode, dialyzer type — Change of hemodialysis mode and dialyzer type

SUMMARY:
Hemodialysis treatment enables patients with end-stage chronic kidney disease to survive. At the same time, however, this treatment also increases cardiovascular mortality, in particular due to a chronically increased level of inflammation and usually incomplete removal of uraemic toxins. Both of these are closely linked with the functional properties of albumin.

The aim of this study is to investigate the effects of various parameters of dialysis, in particular dialyzer properties and dialysis mode on the functional properties of albumin and to what extent these parameters can be used therapeutically, to improve the treatment quality of hemodialysis treatment in the long term by modifying albumin functional properties.

Our own preliminary work in this field and the current state of research indicate that, for example, the use of high-flux dialyzers can contribute to a reduction of the oxidative stress level. It also appears possible that treatment mode (haemodiafiltration instead of haemodialysis) may also have an effect on the binding and detoxification efficiency of albumin and thus on the removal of uraemic toxins.

Previous results have mostly been collected in observational studies. As a proof-of-concept study, this study will further investigate the concrete therapeutic applicability in an interventional study design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at least 3 month of hemodialysis treatment (3x/week) with constant dialysis treatment regimen

Exclusion Criteria:

* Age ≤ 18 years

  * Less than three months of regular (3x/week) hemodialysis treatments or less than 3 treatments/week
  * Acute or chronic liver disease (Child stage A or higher or fulfillment of the of the Kings College criteria)
  * Infusion of commercial human albumin (e.g. in the context of ascites drainage) in the last three months prior to study inclusion
  * Acute or severe chronic infections
  * Acute tumor disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Level of irreversibly oxidized albumin HNA-2 | after 9 month
  change of human mercaptalbumin-2 HNA-2
Level of albumin binding and detoxification efficiency | after 9 month
  Change of albumin binding and detoxification efficiency, meausurement according to PMID: 37558390

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided